CLINICAL TRIAL: NCT05382286
Title: A Randomized, Open-label, Phase 3 Study of Sacituzumab Govitecan and Pembrolizumab Versus Treatment of Physician's Choice and Pembrolizumab in Patients With Previously Untreated, Locally Advanced Inoperable or Metastatic Triple-Negative Breast Cancer, Whose Tumors Express PD-L1
Brief Title: Study of Sacituzumab Govitecan-hziy and Pembrolizumab Versus Treatment of Physician's Choice and Pembrolizumab in Patients With Previously Untreated, Locally Advanced Inoperable or Metastatic Triple-Negative Breast Cancer
Acronym: ASCENT-04
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-592-6173; 2021-005742-14 (EudraCT Number); KEYNOTE-D19 (Other: Merck Sharp & Dohme LLC); jRCT2041220123 (Registry Identifier: Japan Registry of Clinical Trials); MK-3475-D19 (Other: Merck Sharp & Dohme LLC); 2023-504194-21 (Other: European Medicines Agency)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; PD-L1 Positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (SG) + Pembrolizumab (Experimental): Participants will receive SG 10 mg/kg on Days 1 and 8 of 21-day cycles and pembrolizumab 200 mg on Day 1 of 21-day cycles
  Pembrolizumab will be administered for a maximum of 35 cycles.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Pembrolizumab
- Pembrolizumab + Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive pembrolizumab 200 mg on Day 1 of each 21-day cycle (maximum 35 cycles) plus TPC determined prior to randomization from 1 of the 3 allowed regimens:
  * Paclitaxel 90 mg/m^2 on Days 1, 8, and 15 of 28-day cycles
  * nab-Paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of 28-day cycles
  * Gemcitabine 1000 mg/m^2 + carboplatin area under the curve (AUC) 2 on Days 1 and 8 of 21-day cycles
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: nab-Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Sacituzumab Govitecan-hziy (SG) + Pembrolizumab
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
Drug: Paclitaxel — Administered intravenously
  Other Names: Taxol®
  Arms: Pembrolizumab + Treatment of Physician's Choice (TPC)
Drug: nab-Paclitaxel — Administered intravenously
  Other Names: Abraxane®
  Arms: Pembrolizumab + Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — Administered intravenously
  Other Names: Gemzar
  Arms: Pembrolizumab + Treatment of Physician's Choice (TPC)
Drug: Carboplatin — Administered intravenously
  Arms: Pembrolizumab + Treatment of Physician's Choice (TPC)

SUMMARY:
The primary objective of this study is to compare the progression-free survival (PFS) between sacituzumab govitecan-hziy (SG) and pembrolizumab versus treatment of physician's choice (TPC) and pembrolizumab in participants with previously untreated, locally advanced inoperable or metastatic triple-negative breast cancer, whose tumors express programmed cell death ligand 1 (PD-L1).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with locally advanced, inoperable, or metastatic triple-negative breast cancer (TNBC) who have not received previous systemic therapy for advanced disease and whose tumors are programmed cell death ligand 1 (PD-L1) positive at screening.

  * Individuals must have completed treatment for Stage I to III breast cancer, if indicated, and ≥ 6 months must have elapsed between completion of treatment with curative intent and first documented local or distant disease recurrence.
  * Individuals presenting with de novo metastatic TNBC are eligible for this study.
  * TNBC status and tumor PD-L1 combined positive score (CPS) will be confirmed centrally on a recent or archival tumor specimen.
  * Individuals must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria as evaluated locally.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Demonstrates adequate organ function
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Individuals with HIV must be on antiretroviral therapy (ART) and have a well-controlled HIV infection/disease.

Key Exclusion Criteria:

* Positive serum pregnancy test or women who are lactating.
* Received prior therapy with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Individuals may not have received systemic anticancer treatment (with the exception of endocrine therapy) within the previous 6 months or radiation therapy within 2 weeks prior to enrollment.
* Individuals may not be participating in a study with an investigational agent or investigational device within 4 weeks prior to randomization. Individuals participating in observational studies are eligible.
* Have previously received topoisomerase 1 inhibitors or antibody drug conjugates containing a topoisomerase inhibitor.
* Have an active second malignancy.
* Have active serious infection requiring antibiotics.
* Individuals positive for HIV-1 or 2 with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Randomization up to approximately 33 months
  PFS is defined as the time from the date of randomization until the date of objective progressive disease (PD) or death (whichever comes first).

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 53 months
  OS is defined as the time from the date of randomization until death due to any cause.
Objective Response Rate (ORR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 53 months
  ORR is defined as the proportion of participants who achieve complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.
Duration of Response (DOR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 53 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of objective PD or death from any cause (whichever comes first).
Time to Response (TTR) as Assessed by BICR per RECIST Version 1.1 | Randomization up to approximately 53 months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 53 months plus 30 days
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 53 months plus 30 days
Time to Deterioration (TTD) in Global Health Status/Quality of Life (QoL) Scale as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Core Questionnaire, Version 3.0 (EORTC QLQ-C30) | Randomization up to approximately 53 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the participant).
TTD of Pain Score as Measured by EORTC QLQ-C30 | Randomization up to approximately 53 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the participant).
TTD of Fatigue Score as Measured by EORTC QLQ-C30 | Randomization up to approximately 53 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (ie, a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (ie, a worse state of the participant).
TTD of Physical Functioning Domain Score as Measured by EORTC QLQ-C30 | Randomization up to approximately 53 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (ie, a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (ie, a worse state of the participant).
TTD of Role Functioning Score as Measured by EORTC QLQ-C30 | Randomization up to approximately 53 months
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (ie, a better state of the participant), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (ie, a worse state of the participant).

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (504):
- United States (247):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Arizona Oncology Associates, PC-Hope,1845 W Orange Grove Rd, Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope,2070 W. Rudasill Rd., Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope, Tucson, Arizona
  - Arizona Oncology Associates, PC-Hope,1620 West St. Mary's Road, Tucson, Arizona
  - Genesis Cancer and Blood Institute, Hot Springs, Arkansas
  - Genesis Cancer and Blood Institute,1456 Higdon Ferry Road Suite B., Hot Springs, Arkansas
  - Saint Bernards Medical Center, Jonesboro, Arkansas
  - Saint Bernards Medical Center,4000 Linwood Drive, Paragould, Arkansas
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,201 S. Buena Vista Street, Suite 200, Burbank, California
  - University of California Irvine Health Chao Family,1640 Newport Blvd, Costa Mesa, California
  - City of Hope, Duarte, California
  - University of California San Diego Moores Cancer, La Jolla, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,24302 Paseo de Valencia, Suite 200, Laguna Hills, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - City of Hope,1601 Avocado Ave, Newport, California
  - University of California Irvine Health Chao Family, Orange, California
  - City of Hope,209 Fair Oaks Ave, Pasadena, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,892 Aerovista Place, Suite 240, San Luis Obispo, California
  - Sansum Clinic, Santa Barbara, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,2020 Santa Monica Blvd, Suite 600, Santa Monica, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,2336 Santa Monica, Suites 302 and 304, Santa Monica, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Santa Monica, California
  - St. Jude Hospital Yorba dba St. Joseph Heritage Healthcare, Santa Rosa, California
  - Sansum Clinic,2040 Viborg Road, Solvang, California
  - City of Hope,5215 Torrance Blvd, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope,1100 San Bernardino Rd, Upland, California
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center,1250 La Venta Dr, Suite 100, Westlake Village, California
  - Rocky Mountain Cancer Centers,1700 South Potomac Street, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers,2312 N. Nevada Avenue, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers,6031 E. Woodman Rd., Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers,4700 E. Hale Parkway, Denver, Colorado
  - Rocky Mountain Cancer Centers,11750 West 2nd Place, Lakewood, Colorado
  - Rocky Mountain Cancer Centers,22 West Dry Creek Circle, Littleton, Colorado
  - Rocky Mountain Cancer Centers,10107 Ridge Gate Parkway, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers,2030 Mountain View Ave Ste 210, Longmont, Colorado
  - Rocky Mountain Cancer Centers,3676 Parker Blvd, Pueblo, Colorado
  - Rocky Mountain Cancer Centers,525 W. 15th Street, Pueblo, Colorado
  - Rocky Mountain Cancer Centers,8820 Huron Street, Thornton, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Advent Health Medical Group, Altamonte Springs, Florida
  - SCRI - Florida Cancer Specialists - North Region R,750 Orienta Ave, Altamonte Springs, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,2801 NE 213th St, Aventura, Florida
  - Florida Cancer Specialists,9776 Bonita Beach Road Southeast Suite 201 A, Bonita Springs, Florida
  - Florida Cancer Specialists,3630 Manatee Avenue West, Bradenton, Florida
  - Florida Cancer Specialists,5985 Silver Falls Run, Bradenton, Florida
  - SCRI - Florida Cancer Specialists - North Region R,403 S. Kings Ave., Brandon, Florida
  - Florida Cancer Specialists,1030 Commerce Creek Blvd, Cape Coral, Florida
  - SCRI - Florida Cancer Specialists - North Region R,3280 McMullen Booth Road, Clearwater, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,5555 Ponce De Leon Blvd, Coral Gables, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach,224 Memorial Medical Parkway, Suite 300, Daytona Beach, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,1192 East Newport Center Drive, Deerfield Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists,8981 Colonial Center Drive, Fort Myers, Florida
  - Florida Cancer Specialists,8260 Gladiolus Dr, Fort Myers, Florida
  - SCRI - Florida Cancer Specialists - North Region R,6420 W. Newberry Road, Gainesville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,3850 Hollywood Blvd, Hollywood, Florida
  - SCRI - Florida Cancer Specialists - North Region R,100 Highland Avenue, Largo, Florida
  - SCRI - Florida Cancer Specialists - North Region R,521 North Lecanto Highway, Lecanto, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,1400 NW 12th Ave, Miami, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,8932 S.W. 97 Ave, Miami, Florida
  - Florida Cancer Specialists,1100 Goodlette Road, Naples, Florida
  - SCRI - Florida Cancer Specialists - North Region R,4945 SW 49th Place, Ocala, Florida
  - SCRI - Florida Cancer Specialists - North Region R,2824 Enterprise Rd, Orange City, Florida
  - Advent Health Medical Group,2501 North Orange Ave, Orlando, Florida
  - SCRI - Florida Cancer Specialists - North Region R,70 W. Gore Street, Orlando, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center,8100 SW 10 Street, Plantation, Florida
  - Florida Cancer Specialists,22395 Edgewater Drive, Port Charlotte, Florida
  - Florida Cancer Specialists,600 North Cattlemen Road, Sarasota, Florida
  - Florida Cancer Specialists,1970 Golf Street, Sarasota, Florida
  - SCRI - Florida Cancer Specialists - North Region R,7154 Medical Center Drive, Spring Hill, Florida
  - SCRI - Florida Cancer Specialists - North Region R,1201 Fifth Avenue North, St. Petersburg, Florida
  - SCRI - Florida Cancer Specialists - North Region R, St. Petersburg, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach,301 SE Ocean Blvd, Suite 102, Stuart, Florida
  - SCRI - Florida Cancer Specialists - North Region R,3402 West Dr. Martin Luther King Jr. Boulevard, Tampa, Florida
  - SCRI - Florida Cancer Specialists - North Region R,4100 Waterman Way, Tavares, Florida
  - SCRI - Florida Cancer Specialists - North Region R,1400 US Highway 441 N, The Villages, Florida
  - SCRI - Florida Cancer Specialists - North Region R,9320 State Road 54, Trinity, Florida
  - Florida Cancer Specialists,836 Sunset Lake Blvd, Venice, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach,3730 7th Terrace, Suite 101, Vero Beach, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach,1037 S. State Road 7, Bldg B, Suite 303, Wellington, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach, West Palm Beach, Florida
  - SCRI - Florida Cancer Specialists - North Region R,460 N Orlando Ave, Winter Park, Florida
  - Northside Hospital,125 King Avenue, Athens, Georgia
  - Piedmont Cancer Institute - Atlanta,1267 Hwy 54W, Atlanta, Georgia
  - Winship Cancer Institute of Emory University,550 Peachtree St NE, Atlanta, Georgia
  - Piedmont Cancer Institute - Atlanta, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital,5670 Peachtree Dunwoody Rd., Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University,5665 Peachtree Dunwoody Road, Atlanta, Georgia
  - Northside Hospital,308 Deep South Farm Rd, Suite 200, Blairsville, Georgia
  - Northside Hospital,228 Riverstone Dr., Canton, Georgia
  - Northside Hospital,1505 Northside Blvd, Suite 4600, Cumming, Georgia
  - Northside Hospital,3855 Pleasant Hill Rd., Suite 480, Duluth, Georgia
  - Northside Hospital,308 Coliseum Dr., Macon, Georgia
  - Piedmont Cancer Institute - Atlanta,775 Poplar Road, Newnan, Georgia
  - Piedmont Cancer Institute - Atlanta,1240 Eagles Landing Pkwy, Stockbridge, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System (Outpatient Cancer Center), Chicago, Illinois
  - Orchard Healthcare Research Inc,2845 North Sheridan Road, 1st Floor, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,1 Kish Hospital Drive, DeKalb, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,10 Health Services Drive, DeKalb, Illinois
  - Orchard Healthcare Research Inc,800 Austin Street, Suite 360, East Tower, Evanston, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,300 Randall Road, Geneva, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,304 Randall Road, Geneva, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,1000 N. Westmoreland Road, Lake Forest, Illinois
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,4405 Weaver Parkway, Warrenville, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,4455 Weaver Parkway, Warrenville, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University,25 N Winfield Road, Winfield, Illinois
  - Regulatory Management Only: TRIO-US Central Administration, Fort Wayne, Indiana
  - The University of Kansas Cancer Center,2000 Olathe Blvd, Kansas City, Kansas
  - The University of Kansas Cancer Center,12200 W. 110th Street, Overland Park, Kansas
  - The University of Kansas Cancer Center,10710 Nall Avenue, Overland Park, Kansas
  - The University of Kansas Cancer Center,10730 Nall Avenue, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute - Saint Matthews,234 E. Gray Strret, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews,676 S. Floyd Street, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - Norton Cancer Institute - Saint Matthews,4955 Norton Healthcare Blvd, Louisville, Kentucky
  - Hematology Oncology Clinic - Baton Rouge, Baton Rouge, Louisiana
  - Hematology Oncology Clinic - Baton Rouge,1673 E Mount Please Drive, Zachary, Louisiana
  - Cancer Institute Ascension Saint Agnes, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital,102 Endicott Street, Danvers, Massachusetts
  - Massachusetts General Hospital,2014 Washington St, Newton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. John Hospital, Grosse Pointe Woods, Michigan
  - Ascension Providence Hospital Southfield Cancer Center, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The West Clinic, PLLC dba West Cancer Center,7668 Airways Blvd, Southaven, Mississippi
  - The University of Kansas Cancer Center,2750 Clay Edwards Drive, Kansas City, Missouri
  - The University of Kansas Cancer Center,8700 North Green Hills Road, Kansas City, Missouri
  - The University of Kansas Cancer Center,4881 N.E. Goodview Circle, Lee's Summit, Missouri
  - Nebraska Cancer Specialists,2730 W. Faidley Ave, Grand Island, Nebraska
  - Nebraska Cancer Specialists,8303 Dodge Street, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Nebraska Cancer Specialists,611 Fenwick Dr, Papillion, Nebraska
  - Comprehensive Cancer Centers of Nevada - Central V,10001 S. Eastern Avenue, Suite 108, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V,2460 W. Horizon Ridge Parkway, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V,1501 Wigwam Parkway, Suite 1300, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V,653 North Town Center Drive, Suite 402, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V,9280 W. Sunset Road Suite 100, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V,7445 Peak Drive, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central V, Las Vegas, Nevada
  - Summit Medical Group,1 Diamond Hill Road, Berkeley Heights, New Jersey
  - Regional Cancer Care Associates - East Brunswick, East Brunswick, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey,2575 Klockner Road, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey,414 Grand Street, Jersey City, New Jersey
  - Rutgers Cancer Institute of New Jersey,600 River Avenue, Lakewood, New Jersey
  - Rutgers Cancer Institute of New Jersey,94 Old Short Hills Road, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey,300 Second Ave, Long Branch, New Jersey
  - Regional Cancer Care Associates - East Brunswick,9 Centre Drive, Monroe, New Jersey
  - Regional Cancer Care Associates - East Brunswick,34-36 Progress Street, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey,150 Bergen St., Newark, New Jersey
  - Rutgers Cancer Institute of New Jersey,201 Lyons Avenue, Newark, New Jersey
  - Regional Cancer Care Associates - East Brunswick,75 Veronica Avenue, Somerset, New Jersey
  - Rutgers Cancer Institute of New Jersey,110 Rehill Ave, Somerville, New Jersey
  - Rutgers Cancer Institute of New Jersey,99 Highway 37 West, Toms River, New Jersey
  - Rutgers Cancer Institute of New Jersey,100 State Route 36, West Long Branch, New Jersey
  - New York Cancer & Blood Specialists - Port Jeffers,72 East Main St., Babylon, New York
  - Perlmutter Cancer Center - Manhattan - 34th Street,259 First Street, Mineola, New York
  - New York Cancer & Blood Specialists - Port Jeffers,1 Delaware Dr., New Hyde Park, New York
  - Perlmutter Cancer Center - Manhattan - 34th Street, New York, New York
  - NYP/Columbia Univeresity Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - New York Cancer & Blood Specialists - Port Jeffers,365 East Main St., Patchogue, New York
  - New York Cancer & Blood Specialists - Port Jeffers,1500 Rte, 112, Building 4, Port Jefferson, New York
  - New York Cancer & Blood Specialists - Port Jeffers,49 Rte. 347, Newconset Hwy, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Port Jeffers, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Port Jeffers,750 Old County Rd. Suite 4, Riverhead, New York
  - New York Cancer & Blood Specialists - Port Jeffers,12 East 86th St, Suite 4, The Bronx, New York
  - Montefiore Medical Center - Montefiore Medical Park, The Bronx, New York
  - New York Cancer & Blood Specialists - Port Jeffers,2330 Eastchester Road, Suite 360, The Bronx, New York
  - The Ohio State University Wexner Medical Center Clinical Laboratories, Columbus, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Northwest Cancer Specialists, PC,5050 NE Hoyt St., Portland, Oregon
  - Northwest Cancer Specialists, PC,265 N. Broadway, Portland, Oregon
  - Northwest Cancer Specialists, PC, Tigard, Oregon
  - Magee-Womens Hospital of UPMC,200 Oxford Drive, Bethel Park, Pennsylvania
  - Magee-Womens Hospital of UPMC,3 St. Francis Way, Cranberry Township, Pennsylvania
  - Magee-Womens Hospital of UPMC,2500 West 12th Street, Erie, Pennsylvania
  - Magee-Womens Hospital of UPMC,201 State Street, 6 Main, Erie, Pennsylvania
  - Magee-Womens Hospital of UPMC,200 Village Drive, Greensburg, Pennsylvania
  - Magee-Womens Hospital of UPMC,400 Oxford Drive, Monroeville, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC,300 Halket Street, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC,5115 Centre Avenue, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC,9100 Babcock Boulevard, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital of UPMC,100 Fairfield Dr, Seneca, Pennsylvania
  - Magee-Womens Hospital of UPMC,470 Johnson Road, Washington, Pennsylvania
  - Magee-Womens Hospital of UPMC,1703 Innovation Drive, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rhode Island Hospital,164 Summit Ave, Fain 275A, Providence, Rhode Island
  - Tennessee Oncology, PLLC,103 Natchez Park Drive, Dickson, Tennessee
  - Tennessee Oncology, PLLC,4488 Carothers Parkway, Franklin, Tennessee
  - Tennessee Oncology, PLLC,225 Big Station Camp Blvd, Gallatin, Tennessee
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC,353 New Shackle Island Road, Hendersonville, Tennessee
  - Tennessee Oncology, PLLC,5653 First Blvd., Hermitage, Tennessee
  - Tennessee Oncology, PLLC,103 Physicians Way, Lebanon, Tennessee
  - Tennessee Oncology, PLLC,1840 Medical Center Parkway, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC,2004 Hayes Street, Nashville, Tennessee
  - Tennessee Oncology, PLLC,SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC,4220 Harding Rd, Nashville, Tennessee
  - Tennessee Oncology, PLLC,3443 Dickerson Road, Nashville, Tennessee
  - Tennessee Oncology, PLLC,397 Wallace Road, Nashville, Tennessee
  - Tennessee Oncology, PLLC,120 Frank Martin Road, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC,300 Stonecrest Blvd, Smyrna, Tennessee
  - The Center for Cancer and Blood Disorders - Magnolia,515 W. Mayfield Rd., Arlington, Texas
  - Texas Oncology-Austin,901 West 38th Street, Austin, Texas
  - Texas Oncology-Austin, Austin, Texas
  - Texas Oncology-Austin,4101 James Casey, Suite 100, Austin, Texas
  - The Center for Cancer and Blood Disorders - Magnolia,11805 South Freeway, Burleson, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Denison, Denison, Texas
  - The Center for Cancer and Blood Disorders - Magnolia, Fort Worth, Texas
  - Oncology Consultants,1631 North Loop West, Houston, Texas
  - Oncology Consultants,925 Gessner, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - University of Texas MD Anderson Cancer Center,1155 Pressler St, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - The Center for Cancer and Blood Disorders - Magnolia,920 Santa Fe Drive, Weatherford, Texas
  - Huntsman Cancer Institute, University of Utah,165 North University Avenue, Farmington, Utah
  - Huntsman Cancer Institute, University of Utah,1280 E. Stringham Avenue, Salt Lake City, Utah
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Huntsman Cancer Institute, University of Utah,5126 West Daybreak Parkway, South Jordan, Utah
  - Virginia Oncology Associates,744 N. Battlefield Blvd, Chesapeake, Virginia
  - Virginia Cancer Institute,7501 Right Flank Road, Mechanicsville, Virginia
  - Virginia Oncology Associates,1051 Loftis Blvd Suite 100, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute,210 Medical Park Boulevard, Petersburg, Virginia
  - Virginia Cancer Institute,1401 Johnston-Willis Drive, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Oncology Associates,1950 Glenn Mitchell Drive, Virginia Beach, Virginia
  - Northwest Cancer Specialists, PC,210 SE 136th Avenue, Vancouver, Washington
- Argentina (6):
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Instituto de Oncología Ángel H. Roffo, CABA
  - Fundacion CORI para la Investigacioy y Prevención del Cancer, Capital
  - Instituto de Oncologia de Rosario, Rosario
  - CAIPO Centro Para La Atención Integral Del Pacient, San Miguel de Tucumán
  - Clinica Viedma, Viedma
- Australia (12):
  - Border Medical Oncology, Albury, New South Wales
  - Saint George Hospital - Australia, Kogarah, New South Wales
  - Mater Hospital - North Sydney, North Sydney, New South Wales
  - GenesisCare - North Shore, St Leonards, New South Wales
  - Mater Misericordiae Limited and Mater Research Limited, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Cancer Research SA (CRSA), Adelaide, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - Breast Cancer Research Center - Western Australia, Nedlands, Western Australia
- Austria (5):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitätsklinikum Sankt Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
- Belgium (8):
  - Institut Jules Bordet, Anderlecht
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Grand Hopital de Charleroi - Notre Dame, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire Université Cathol, Namur
- Brazil (14):
  - Hospital Araújo Jorge - Associacao de Combate ao Cancer em Goias - ACCG, Goiânia
  - Centro de Pesquisa Clinica Em Oncologia - ONCOSITE, Ijuí
  - Hospital de Clinicas de Porto Alegre - HCPA, Itajaí
  - Centro de Pesquisas Clinicas da Fundacao Doutor Amaral Carvalho - Hospital Amarval Carvalho, Jaú
  - Associacao Hosptialar Moinos de Vento - Hospital Moinhos de Vento, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto Nacional de Câncer - Brazil, Rio de Janeiro
  - Núcleo de Oncologia da Bahia, Salvador
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia - Centro Universitário FMABC, Santo André
  - Real e Benemerita Associacao Portuguesa de Beneficencia - Hospital Beneficencia Portuguesa (BP) - Unidade Paulista, São Paulo
  - Clinica de Pesquisas e Centro de Estudos em Oncolo, São Paulo
  - Fundação Pio XII - Hospital de Câncer de Barretos, São Paulo
  - Nucleo de Pesquisa Clinica da Rede Sao Camilo, São Paulo
- Canada (12):
  - Tom Baker Cancer Centre, Calgary
  - Cross Cancer Institute, Edmonton
  - QEII Health Sciences Centre, Halifax
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener
  - London Health Sciences Centre, London
  - Jewish General Hospital, Montreal
  - McGill University Health Centre, Montreal
  - Princess Margaret Cancer Centre - University Health Network, Ontario
  - Ottawa Hospital - General Campus, Ottawa
  - Sunnybrook Research Institute, Toronto
  - Mount Sinai Hospital, Toronto
  - British Columbia Cancer - Vancouver, Vancouver
- Chile (5):
  - Oncovida - Santiago, Providencia
  - Clínica Alemana, Santiago
  - Clínica IRAM, Santiago
  - Centro de Cancer Pontificia Universidad Catolica, Santiago Region
  - James Lind Centro de Investigacion del Cancer, Temuco
- Czechia (6):
  - Masarykuv Onkologicky Ustav, Klinika Komplexni Onkologicke Pece, Brno
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní Thomayerova nemocnice, Hradec Králové
  - Fakultni nemocnice Olomouc, Onkologicka klinika, Olomouc
  - Fakultní Nemocnice Královské Vinohrady, Radioterapeuticka a onkologicka klinika, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Onkologicka klinika, Prague
- France (16):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Centre Hospitalier Régional et Universitaire de Be, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital Morvan, Institut de cancérologie, Brest
  - Centre de Lutte contre le Cancer - François Bacles, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Hospices Civils de Lyon, Hôpital Lyon Sud, Pierre-Bénite
  - Centre Armoricain de Radiothérapie, dImagerie Méd, Plérin
  - Centre Eugène Marquis, Rennes
  - Institut Claudius Regaud - IUCT-O, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (18):
  - Helios Klinikum Berlin-Buch, Berlin
  - : Gynakologisches Zentrum Bonn, Schwerpunkt Gyn. Onkologie,, Bonn
  - Marienhospital Bottrop, Bottrop
  - Klinik Frauenheilkunde, Uniklinik ClO, Studienzentrale, Cologne
  - Universitätsklinikum Erlangen, Frauen klinik, Erlangen
  - Kliniken Essen-Mitte - Evangelische Huyssens-Stift, Essen
  - Praxis für interdisziplinäre Onkologie & Hämatolog, Freiburg im Breisgau
  - : Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Facharztzentrum Eppendorf, Hamburg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universitätsklinikum Schleswig-Holstein Institut fur Klinische Chermie, Lübeck
  - Universitatsklinikum Mannheim GmBH, Frauenklinik, Mannheim
  - EV. Krankenhaus Bethesda - Johanniter GmbH, Station 1 Brustzentrum Niederrhein, Mönchengladbach
  - Rotkreuzklinikum Munchen Frauenklinik, München
  - Klinik und Poliklinik für Frauenheilkunde, München
  - Universitätsklinikum Münster, Bereich Senologie an der klinik fur Frauenheilkunde und Gerburtschilfe, Münster
  - Universitatsklinikum Tubingen, Tübingen
  - St. Josefs-Hospital Wiesbaden GmbH, Gynakologie und Geburtshilfe, Wiesbaden
- Hong Kong (4):
  - Department of Medicine, Queen Mary Hospital, Hong Kong
  - Hong Kong Sanatorium and Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital - Hong Kong, New Territories
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Petz Aladár Egyetemi Oktató Kórház - Gy?r, Győr
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah - Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center Hospital - Tel Hashomer, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (19):
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - SSD Oncologia Medica Addarii-Zamagni, IRCSS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - UO Oncologia, ASST degli Spedali Civili di Brescia, Brescia
  - IRCCS Ospedale Policlinico San Martino, Genova GE
  - S.C. Oncologia medica, ASST di Lecco, Lecco
  - Presidio Ospedaliero di Lucca, Lucca
  - Ospedale Generale Provinciale - Macerata, Macerata
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Centro Ricerca Fase I, Fondazione IRCSS San Gerado dei Tintori, Monza
  - AOU "Luigi Vanvitelli", Napoli
  - Oncologia Medica Senologica Sperimentale - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - AOU Maggiore della Carita, Novara
  - Istituto Oncologico Veneto - IRCCS, Padua
  - S.O.C Oncologia Medica, Nuovo Ospedale di Prato Santo Stefano, Prato
  - Policlinico di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Geme, Rome
  - Azienda Ospedaliera Universitaria Senese - Losped, Siena
- Japan (28):
  - Aichi Cancer Center Hospital, Aichi
  - Tohoku University Hospital, Aoba-ku
  - Juntendo University Hospital, Bunkyō City
  - Chiba Cancer Center, Chūōku
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Chūōku
  - NHO Shikoku Cancer Center, Ehime
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Cancer Center, Inamachi
  - Hakuaikai Sagara Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Kumamoto University Hospital, Kumamoto
  - Kure Medical Center And Chugoku Cancer Center, Kure
  - Mie University Hospital, Mie
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Hiroshima City Hiroshima Citizens Hospital, Nakaku
  - NIigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Kyoto University Hospital, Sakyo-ku
  - Hokkaido Cancer Center, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Showa University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Malaysia (8):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
  - Institut Kanser Negara, Putrajaya
  - Hospital Wanita dan Kanak-Kanak Sabah, Sabak Bernam
  - Sarawak General Hospital, Sarawak
- Mexico (10):
  - Icaro Investigaciones en Medicina S.A. de C.V., Chihuahua City
  - Centro para el Desarrollo de la Medicina, Culiacán
  - Panamerican Clinical Research Mexico - Guadalajara, Guadalajara
  - Cryptex Investigación Clínica, Mexico City
  - Medical Care and Research S.A. de C.V, Mérida
  - Fucam A.C., México
  - Avix Investigacion Clinica S.C., Monterrey
  - Oncológico Potosino, San Luis Potosí City
  - FAICIC Clínical Research, Veracruz
  - iBiomed - Investigacion Biomedica para el Desarrol, Zapopan
- Netherlands (4):
  - Amphia Ziekenhuis - Breda Langendijk, Breda
  - Universitair Medisch Centrum Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus Medisch Centrum, Rotterdam
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej, Gliwice
  - SP ZOZ Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego, Opole
  - Wielkopolskie Centrum Onkologii im. Marii Sklodowskiej-Curie, Poznan
  - Mazowiecki Szpital Wojewódzki im. w. Jana Pawa II w, Siedlce
  - Narodowy Instytut Onkologii im.Marii Marii Sklodowskiejs, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Ponce Medical School Foundation Inc., Ponce, PR, Puerto Rico
- South Africa (3):
  - Hopelands Cancer Centre, Hilton
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - University of Pretoria, Pretoria
- South Korea (8):
  - National Cancer Center - Korea, Goyang-si Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (17):
  - Hospital Teresa Herrera - Materno Infantil, A Coruña
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Centre Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Unviersitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- Switzerland (5):
  - Kantonsspital Baden, Baden
  - Kantonsspital Baselland - Standort Liestal, Liestal
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Brust-Zentrum Zurich, Zurich
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (12):
  - Baskent Uni. Dr Turgut Noyan Uyg. ve Aras. Merkezi, Adana
  - Ankara Il Saglik Mudurlugu SBU Gulhane Egitim Ve A, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Hacettepe Üniversitesi Hastanesi, Ankara
  - Trakya Universitesi Tip Fakultesi Hastanesi, Edirne
  - Istanbul Il Saglik Mudurlugu Goztepe Prof. Dr. Sul, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - Medicana International Izmir Hastanesi, Izmir
  - Acibadem Maslak Hastanesi, Sarıyer
  - VKV Amerikan Hastanesi, Şişli
- United Kingdom (8):
  - NHS Lothian, Edinburgh
  - Clinical Trials Unit Lvl 0 Cancer Research UK Beatson Institute, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - : Barts Health NHS Trust, St Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Guy's and Saint Thomas' NHS Foundation Trust, London
  - University College London Hospitals, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolaney SM, de Azambuja E, Kalinsky K, Loi S, Kim SB, Yam C, Rapoport B, Im SA, Pistilli B, Mchayleh W, Cescon DW, Watanabe J, Banuelas MAL, Freitas-Junior R, Salvador Bofill J, Afshari M, Gary D, Wang L, Lai C, Schmid P; ASCENT-04/KEYNOTE-D19 Clinical Trial Investigators. Sacituzumab Govitecan plus Pembrolizumab for Advanced Triple-Negative Breast Cancer. N Engl J Med. 2026 Jan 22;394(4):354-366. doi: 10.1056/NEJMoa2508959. PMID 41564397
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-592-6173